CLINICAL TRIAL: NCT05107414
Title: Multi-center In Vivo Kinematics for Subjects Implanted With Smith & Nephew Journey II BCS TKA, Journey II CR TKA, Or Journey II XR TKA
Brief Title: Journey 2 Multi Center Kinematic Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Sponsor
Other Study IDs: 20203268
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2023-05

CONDITIONS: Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (3):
- Journey II Bi-Cruciate Stabilized: Participants who have been implanted with a Smith & Nephew Journey II BCS TKA
  Interventions: Procedure: Total Knee Arthroplasty
- Journey II Cruciate Retaining: Participants who have been implanted with a Smith & Nephew Journey II CR TKA
  Interventions: Procedure: Total Knee Arthroplasty
- Journey II Bi-Cruciate Retaining: Participants who have been implanted with a Smith & Nephew Journey II BCR TKA
  Interventions: Procedure: Total Knee Arthroplasty

INTERVENTIONS:
Procedure: Total Knee Arthroplasty — Participants have previously undergone a total knee replacement surgery.
  Other Names: Smith & Nephew Journey II TKA

SUMMARY:
The objective of this study is to determine and compare the in vivo kinematics and vibroarthrography (VAG) signals for subjects implanted with Journey II Bi-Cruciate Stabilized (BCS), CR (Cruciate Retaining), and Bi-Cruciate Retaining (XR) TKAs.

ELIGIBILITY:
Inclusion Criteria:

1. Patients in the age range of 18 years to 85 years (both inclusive)
2. Patients who have a BMI less than 35
3. Patients who do not have previous surgery on the implanted knee that might restrict their movement
4. Patient who are at least 6 months post-operative
5. Patients who do not experience any pain or other post-operative complications
6. Patients who have a stable TKA and can perform a deep knee bend activity
7. Patients who are willing to participate in this study and are willing to sign appropriate HIPAA and informed consent forms
8. Subjects will have a Journey II knee system

Exclusion Criteria:

1. Pregnant, potentially pregnant, or lactating females. To satisfy radiation protocol, each female subject will be asked if she is pregnant, or possibly could be pregnant. A pregnant person will not be allowed to participate in the study.
2. Patients who have currently enrolled in a fluoroscopic study within the past year.
3. Patients currently involved in any personal injury litigation, medical/legal or workman's compensation claims.
4. Patients with known drug or alcohol abuse histories or psychological disorders that could affect ability to complete all aspects of the study.
5. Patients with neurological or musculoskeletal disorders that might adversely affect weight-bearing motion ability
6. Subjects who are unable to perform a deep knee bend.
7. Subjects who are unwilling to sign Informed Consent/ HIPAA documents.
8. Subjects without the required type of knee implant.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All participants will be selected by their respective surgeons. Participants will be screened by eligible surgeon staff and will have the required implant for each site.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Estimated)
Dates: Start 2021-05-15 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Femorotibial Medial Condylar Rollback | Baseline, at time of observation
  The condylar rollback of the medial condyle will be observed at a single instance in time. Participants will have previously undergone a total knee arthroplasty but data cannot be collected on their preoperative kinematics. Outcome will be measured in [mm].
Femorotibial Lateral Condylar Rollback | Baseline, at time of observation
  The condylar rollback of the lateral condyle will be observed at a single instance in time. Participants will have previously undergone a total knee arthroplasty but data cannot be collected on their preoperative kinematics. Outcome will be measured in [mm].
Femorotibial Axial Rotation | Baseline, at time of observation
  The femorotibial axial rotation will be observed at a single instance in time. Participants will have previously undergone a total knee arthroplasty but data cannot be collected on their preoperative kinematics. Outcome will be measured in [deg].
Femorotibial Weight Bearing Flexion | Baseline, at time of observation
  The femorotibial weight bearing flexion will be observed at a single instance in time. Participants will have previously undergone a total knee arthroplasty but data cannot be collected on their preoperative kinematics. Outcome will be measured in [deg].

CONTACTS AND LOCATIONS:
Locations (1):
- University of Tennessee, Knoxville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No